CLINICAL TRIAL: NCT00153400
Title: The California Well-Integrated Screening and Evaluation for Women Across the Nation (WISEWOMAN) Project: Improving Cardiovascular Risk Factors for Underserved Hispanic Women
Brief Title: The California WISEWOMAN Project:Cardiovascular(CVD) Health for Hispanic Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of California, San Francisco (Other); California Department of Health Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDC-NCCDPHP-3898; U58/CCU922827-01 (Other Grant/Funding Number: Centers for Disease Control and Prevention)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Cardiovascular Diseases; Chronic Diseases
Keywords: CVD risk
MeSH Terms: conditions — Cardiovascular Diseases; Chronic Disease | interventions — Walking; methyl hydroxyethyl cellulose

STUDY DESIGN:
Intervention Model Description: Provide Health coaching and Lifestyle programs
Masking Description: Low income uninsured and underinsured participants.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Enhanced Lifestyle Intervention (Experimental): Three health coaching sessions or Lifestyle Programs on physical activity and nutrition are delivered to each woman. Support is offered by community health workers.
  Interventions: Behavioral: Enhanced Lifestyle Intervention

INTERVENTIONS:
Behavioral: Enhanced Lifestyle Intervention — Three face-to-face counseling sessions for nutrition and physical activity. Used a Spanish culturally tailored materials. These interventions were delivered by community health workers (CHWs) who are trained.
  Other Names: YWCA Health Coaching and Walk with Ease

SUMMARY:
The purpose of this trial is to provide low-income, under- or un-insured 40- to 64-year-old women with the knowledge, skills, and opportunities to improve diet, physical activity, and other lifestyle behaviors to prevent, delay and control cardiovascular and other chronic diseases.

DETAILED DESCRIPTION:
This study is based on a single group. Evaluated how effectively culturally appropriate lifestyle intervention was in improving, over a relatively short-term period (~12 months) on health behaviors and the CVD risk profile.

ELIGIBILITY:
Inclusion Criteria:

* National Breast and Cervical Cancer Early Detection Program (NBCCEDP)participants without cancer
* Income < 200 percent of federal poverty level
* Under or uninsured for the health care coverage
* Blood pressure >= 120 mm Hg systolic or >=80 mm Hg diastolic or currently taking medication to lower cholesterol

Exclusion Criteria:

* >180 mm Hg systolic or >110 mm Hg diastolic
* > 400 cholesterol
* pregnant women
* had past or current CVD events

Ages: 40 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2006-01; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
CVD risk (10 year estimated risk) | baseline, one-year
  Combines a number of risk factors into one metric. Lower score means lower risk. Higher score means higher risk. Low risk (0 to <5, borderline risk (5 to <7.5), intermediate risk (7.5 to < 20), and high risk (>20). Range 0 to 20.

SECONDARY OUTCOMES:
Physical Activity | baseline, one-year
  Number of minutes of physical activity per week. American Heart Association recommendation of 150 mins per week for good health. Self-recorded daily and self-reported weekly.
Dietary Behavior | baseline, one-year
  Numbers of fruits and vegetables on a weekly basis. The NHLBI standard of measurement is 5-a-day. Self-recorded daily and self-reported weekly.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Will, Study Chair — Centers for Disease Control and Prevention

REFERENCES:
- [Background] Silverstein RP, VanderVos M, Welch H, Long A, Kabore CD, Hootman JM. Self-Directed Walk With Ease Workplace Wellness Program - Montana, 2015-2017. MMWR Morb Mortal Wkly Rep. 2018 Nov 23;67(46):1295-1299. doi: 10.15585/mmwr.mm6746a3. PMID 30462629
- [Result] Ahmann E, Saviet M, Conboy L, Smith K, Iachini B, DeMartin R. Health and Wellness Coaching and Sustained Gains: A Rapid Systematic Review. Am J Lifestyle Med. 2023 Jun 20;18(2):162-180. doi: 10.1177/15598276231180117. eCollection 2024 Mar-Apr. PMID 38559782